CLINICAL TRIAL: NCT04312685
Title: Transitioning to a Valve -Gated Intrathecal Drug Delivery System (IDDS): An Open-Label, Non-Randomized, Single-Blind, Multi-Center Study
Brief Title: Transitioning to a Valve -Gated Intrathecal Drug Delivery System
Acronym: TRANSIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Bux, Anjum, MD (Other)
Collaborators: Flowonix Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T-001
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Pain; Pain, Chronic; Pain, Intractable; Pain, Back
Keywords: IDDS; Intrathecal drug therapy; pain pump
MeSH Terms: conditions — Pain; Chronic Pain; Pain, Intractable; Back Pain

STUDY DESIGN:
Intervention Model Description: Open-Label, Non-Randomized, Single-Blind, Multi-Center
Who Masked: Participant
Masking Description: subject will be blinded to dosing decreases and increases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Prometra Programmable Pump (Active Comparator): Pain scores and drug doses will be prospectively collected for valve-gated Prometra® Programmable Pump system(Flowonix Medical)' at (refills 1-3) and will be compared to 3 months retrospectively collected pain scores (VAS, ODI and Global Pain Scale Assessments) and drug doses prior to peristaltic pump explant.
  Interventions: Device: Prometra II Programmable Pump system - Flowonix Medical
- Retrospective records for peristaltic pump (No Intervention): Prior pain scores and drug doses from the patients who need a new valve gated pump will be recorded and used for comparison after it is changed.

INTERVENTIONS:
Device: Prometra II Programmable Pump system - Flowonix Medical — This valve gated Prometra II Programmable Pump system will be replacing prior peristaltic Synchromed II pump
  Other Names: Prior peristaltic Synchromed II pump
  Arms: Prometra Programmable Pump

SUMMARY:
This study is designed to explore if the valve-gated pump requires less drug to manage subject pain than the prior standard peristaltic pump in the same subject. The newly implanted valve-gated pump will be programmed to deliver a minimum dose reduction of 20% of the same medication that was delivered in the peristaltic pump prior to explant. The drug therapy will be evaluated and pain scores will be evaluated over time (3 refill cycles prospectively for the valve-gated pump and 6 months retrospectively for the peristaltic pump).

DETAILED DESCRIPTION:
This study will employ a single-blind where study participants will not be told about the dose reduction of at least 20% when the valve-gated pump is implanted. A study participant has a significant potential to bias when informed they will get less drug with the new pump than they were receiving in the old pump this could subjectively affect pain scores as well. After valve-gated pump implant and dose reduction, the appropriate pain therapy will be provided to adequately address pain management in the opinion of the study investigator using standard of care processes and VAS scores.

Once subjects have been implanted with the valve-gated pump they will be started on a minimum 20% dose reduction (same medications and concentrations prior to explant). If at any time during the subjects' treatment it is determined by the investigator that the subjects' treatment dose needs to be increased, the dose can be increased in increments not to exceed 5% (no change to concentration) based on VAS scores at current and last visits.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria will be eligible for enrollment in the study:

* 21 years of age or older
* Provide written informed consent for study participation
* Active existing peristaltic intrathecal drug delivery system (IDDS)
* Stable IDDS dosage and concentration for at least 6 weeks prior to valve-gated pump implant
* Minimum of 3 months of information from the following:
* VAS, ODI, Global Pain Scale
* Pump refill printouts (dosage and concentration)
* Other Interventions for pain (injections, nerve blocks, etc.)
* Estimated Replacement Indicator (ERI) printout required showing < 12 months of battery life
* Catheter Access Procedure (CAP) study performed to document patency of catheter, if not replacing
* Diagnosis of nonmalignant, chronic intractable pain as documented in medical history
* Appropriate candidate for surgery
* Able to comply with study requirements including visits and assessments, in the opinion of the investigator

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from participating in the study:

* Any contraindications listed in the Prometra labeling
* Significant pain disorder not intended to be treated with the test device or comparator
* Terminally ill, malignant cancer diagnosis and/or has a life expectancy of less than 12 months in the opinion of the investigator
* Pregnant/lactating woman or is of child-bearing potential and not utilizing effective birth control.
* Systemic or local infection (contraindicated for pump implantation)
* History/evidence of an active disruptive psychiatric disorder or other known condition with potential to impact compliance with study visits and assessments, in the investigator's opinion

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Reduced pain medication through Prometra Implantable Pump System | 12 months
  Total consumption of pain medications both oral and intrathecal is recorded to show changes.

SECONDARY OUTCOMES:
Visual Analog Scale for Pain changes | 12 months
  Visual Analog Scale (VAS) for Pain is used assess pain throughout the study which shows No pain at low end to extreme Pain at high end.
Owestry Disability Index changes | 12 months
  Owestry Disability Index (ODI) are used to assess changes in lifestyle scores throughout the study which shows patient's level of function in daily living
Global Pain Scale Assessments | 12 months
  Global Pain Scale Assessments will be used to assess changes in scores throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Anjum Bux, MD, Principal Investigator — Owner
Locations (8):
- United States (8):
  - Pain and Spine Specialists, Idaho Falls, Idaho
  - Crimson Pain Management, Overland Park, Kansas
  - Bux Pain Management, Lexington, Kentucky
  - Aust Interventional Pain, Slidell, Louisiana
  - Michigan Head & Spine Institute, Southfield, Michigan
  - National Spine & Pain Center, Turnersville, New Jersey
  - The Spine Center at Ridgeway, Rochester, New York
  - Consultants in Pain Management, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knight KH, Brand FM, Mchaourab AS, Veneziano G. Implantable intrathecal pumps for chronic pain: highlights and updates. Croat Med J. 2007 Feb;48(1):22-34. PMID 17309136
- [Background] Deer TR, Smith HS, Cousins M, Doleys DM, Levy RM, Rathmell JP, Staats PS, Wallace M, Webster LR. Consensus guidelines for the selection and implantation of patients with noncancer pain for intrathecal drug delivery. Pain Physician. 2010 May-Jun;13(3):E175-213. PMID 20495597
- [Background] Hayek SM, Deer TR, Pope JE, Panchal SJ, Patel VB. Intrathecal therapy for cancer and non-cancer pain. Pain Physician. 2011 May-Jun;14(3):219-48. PMID 21587327
- [Background] Hayek SM, Veizi E, Hanes M. Intrathecal Hydromorphone and Bupivacaine Combination Therapy for Post-Laminectomy Syndrome Optimized with Patient-Activated Bolus Device. Pain Med. 2016 Mar;17(3):561-571. doi: 10.1093/pm/pnv021. Epub 2015 Dec 14. PMID 26814257
- [Background] Konrad PE, Huffman JM, Stearns LM, Plunkett RJ, Grigsby EJ, Stromberg EK, Roediger MP, Wells MD, Weaver TW. Intrathecal Drug Delivery Systems (IDDS): The Implantable Systems Performance Registry (ISPR). Neuromodulation. 2016 Dec;19(8):848-856. doi: 10.1111/ner.12524. Epub 2016 Oct 12. PMID 27730704
- [Background] Tangen KM, Leval R, Mehta AI, Linninger AA. Computational and In Vitro Experimental Investigation of Intrathecal Drug Distribution: Parametric Study of the Effect of Injection Volume, Cerebrospinal Fluid Pulsatility, and Drug Uptake. Anesth Analg. 2017 May;124(5):1686-1696. doi: 10.1213/ANE.0000000000002011. PMID 28431428